CLINICAL TRIAL: NCT03833856
Title: Incidence and Risk of Poor Outcomes After Colonoscopy Related Perforation: Result From a Prospective Data Registry
Brief Title: Incidence and Clinical Course of Colonoscopy Related Perforation
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Professor, Kyungpook National University Hospital
Other Study IDs: KNUH2019
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Perforation Colon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: colonoscopy perforation — The development of perforation after colonoscopy

SUMMARY:
This study aims to investigate the incidence and clinical course of colonoscopy related perforation based on the result of a prospective registry.

DETAILED DESCRIPTION:
In each endoscopy unit from participating hospital, there is a alarm system focusing on the development of perforation. Therefore, perforation cases will not be missed from the registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a perforation after colonoscopy

Exclusion Criteria:

* Patients who refuse to be registered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients undergoing colonoscopy who end up with perforation.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Operation | 1 month
  Number of participants who take surgical treatment after perforation

CONTACTS AND LOCATIONS:
Overall Officials: Eun Soo Kim, MD, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No